CLINICAL TRIAL: NCT05162599
Title: Evaluation of Cardiags Trimod, a New Medical Device for Screening Cardiac Abnormalities
Brief Title: Evaluation of Cardiags Trimod for Analysis of Cardiac Activity
Acronym: EVALTRIMOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CARDIAGS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDGS-EC-01
Record Dates: First submitted 2021-12-06; First posted 2021-12-17 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-06

CONDITIONS: Murmur, Heart; Rhythm; Abnormal
Keywords: Medical examination device; Connected cardiac auscultation; Sensors; Heartbeat; Heart sounds; Pulse wave; Electrocardiogram; Pathological heart sounds
MeSH Terms: conditions — Heart Murmurs; Arrhythmias, Cardiac | interventions — Diagnostic Techniques and Procedures

STUDY DESIGN:
Intervention Model Description: This is a cross-sectional diagnostic study with collection of information from the gold standard (or reference tests) and the new device
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic study, experimental evaluative cross-sectional study (Experimental): Evaluate the performance of the Cardiags Trimod medical device, compared to a reference examination, echocardiography, for the detection of heart murmurs Verification of the performance of the Cardiags Trimod medical device compared to a reference examination (ECG, Cardiologist interpretation) for the detection of rythm abnormalities Verification of the repeatability of measurements Verification of safety and suitability for use Verification of acceptability
  Interventions: Device: Diagnostic study, experimental evaluative cross-sectional study

INTERVENTIONS:
Device: Diagnostic study, experimental evaluative cross-sectional study — This is a cross-sectional diagnostic study with collection of information from the gold standard (or reference test) and the new device
  Other Names: Noinvasive multisensors cardiac examination

SUMMARY:
The current study concerns Cardiags Trimod, a new non-invasive medical device for cardiac examinations. The evaluation of its effectiveness is done relative to specific standard devices.

DETAILED DESCRIPTION:
Cardiags Trimod, the subject of this study, is a new medical device for rapid and early detection of some of cardiac abnormalities, easy to use by non-cardiologists and portable wherever the patient is. Cardiags Trimod, consisting of a device and software, allows simultaneous recording, visualization and analysis in real time of signals characteristic of cardiac function. It assists healthcare professionals by measuring characteristic time intervals of cardiac function by crossing the various signals, by detecting abnormal rhythms, and murmurs.

The study aims to assess the essential requirements : the effectiveness and safety of the device. The study is a research involving the human person.Cardiags Trimod is a medical device with low risk. There is no identified risk for the patient.The patient sample tested consists of sick and healthy individuals. The use of Cardiags Trimod is part of the patient's usual consultation. The identified Gold standards are EKG and echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Persons suitable for receiving an echocardiogram and an electrocardiogram,
* People who signed the consent form,

Exclusion Criteria:

* Protected and vulnerable people,
* People refusing to participate in the study,

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Murmurs detection | 15 minutes
  Evaluate the performance of Cardiags Trimod compared to a reference examination, echocardiography, for the detection of murmurs: Presence/Absence
Heart rhythm disorders | 15 minutes
  Abnormal and irregular heart rhythm

SECONDARY OUTCOMES:
Accuracy of cardiac intervals measures | 15 minutes
  Measures accuracy
Reproductibilty of measurements | 15 minutes
  Repetition of three measurements by the same operator
Security and usability | 1 year
  collection of problems and incidents during clinical study
Acceptability | 1 year
  satisfaction survey

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Mr Boisson, Dr, Principal Investigator — Hopital Fourvière Lyon France; Bernard Mr RITZ, Dr, Principal Investigator — Hopital Fourvière Lyon France
Locations (1):
- Hôpital de Fourvière, Lyon, France

IPD SHARING:
Plan to Share IPD: No